CLINICAL TRIAL: NCT01791842
Title: TREATMENT OF FIBROUS DYSPLASIA OF BONE WITH TOCILIZUMAB AMONG PATIENTS WHO DO NOT RESPOND TO BISPHOSPHONATES. THE TOCIDYS TRIAL.
Brief Title: TOCILIZUMAB IN FIBROUS DYSPLASIA OF BONE
Acronym: TOCIDYS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010.648; 2010-024282-41 (EudraCT Number)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fibrous Dysplasia of Bone
Keywords: fibrous dysplasia of bone; tocilizumab; McCune-Albright syndrome
MeSH Terms: conditions — Fibrous Dysplasia of Bone; Fibrous Dysplasia, Polyostotic | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tocilizumab first, then placebo (Experimental): one IV infusion per month of Tocilizumab for 6 months followed by 1 infusion per month of placebo, for 6 months.
  Interventions: Drug: Tocilizumab; Drug: Placebo
- Placebo first, then Tocilizumab (Experimental): one IV infusion per month of Placebo for 6 months followed by 1 infusion per month of Tocilizumab, for 6 months.
  Interventions: Drug: Tocilizumab; Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab — 8 mg/kg/month
Drug: Placebo

SUMMARY:
Bone pain due to fibrous dysplasia of bone is usually treated with bisphosphonates. A small proportion of patients fail to respond adequately. Mutated bone cells produce large amounts of Interleukin-6 (IL-6), with increased bone resorption as a result. Inhibition of IL-6 may be of interest to reduce bone resorption and therefore bone pain. TOCIDYS is a placebo-controlled randomized cross-over trial to test the hypothesis that tocilizumab can reduce bone resorption in those patients with fibrous dysplasia who have already received bisphosphonates.

ELIGIBILITY:
Inclusion Criteria:

* fibrous dysplasia of bone
* previously treated with IV bisphosphonates
* persistent bone pain and increased bone remodeling

Exclusion Criteria:

* Chronic renal failure
* serious infectious diseases
* liver enzymes abnormality
* pregnancy
* dyslipidemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-05-05 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
serum CTX (type 1 collagen C-terminal breakdown product) | 6 months

SECONDARY OUTCOMES:
Bone pain | 6 months
  visual analog scale
serum ICTP (Carboxyterminal Telopeptide of Type I Collagen) | 6 months
bone alkaline phosphatase | 6 months
radiographs of mostly affected area | 12 months

OTHER OUTCOMES:
Biological safety | 12 months
  serum creatinine level, red blood cells, white blood cells, platelets, ASAT (Aspartate Amino Transferase), ALAT (Alanine Amino Transferase), CRP (C Reactive Protein) : each month cholesterol, triglycerides : before experimental treatment administration and at 8 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de Rhumatologie, Groupe Hospitalier Pellegrin, Bordeaux
  - Service de rhumatologie, Hopital Edouard Herriot, HCL, Lyon
  - Service de rhumatologie, Hôpital Lariboisière, Paris

REFERENCES:
- [Background] Chapurlat R, Gensburger D, Trolliet C, Rouanet S, Mehsen-Cetre N, Orcel P. Inhibition of IL-6 in the treatment of fibrous dysplasia of bone: The randomized double-blind placebo-controlled TOCIDYS trial. Bone. 2022 Apr;157:116343. doi: 10.1016/j.bone.2022.116343. Epub 2022 Jan 29. PMID 35104665
- See also: Related Info — http://www.dysplasie-fibreuse-des-os.info